CLINICAL TRIAL: NCT02372838
Title: Reconstruction of Extensive Upper Extremity Long Bone Defects With a Microvascular Fibula Flap: a Cross-sectional Study of Long-term Outcomes
Brief Title: Reconstruction of Extensive Upper Extremity Long Bone Defects With a Microvascular Fibula Flap
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jussi Repo, M.S., Helsinki University Central Hospital
Other Study IDs: 343/13/03/02/13/3
Record Dates: First submitted 2015-02-21; First posted 2015-02-26 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Limb Salvage

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Microvascular fibula bone transfer — Reconstructive surgery with a microvascular bone flap

SUMMARY:
This study assesses the long-term functional outcomes of upper extremity long bone defects treated with the free fibula bone transfer.

DETAILED DESCRIPTION:
The study design entails a retrospective review of hospital records and a cross-sectional assessment using patient-reported outcome measures. The purpose of this study is to evaluate the reliability, complications and flap survival rate as well as the long-term functional and health-related quality of life results in patients with upper extremity long bone defect reconstructed using a microvascular fibula bone transfer.

ELIGIBILITY:
Inclusion Criteria:

* All patients of upper extremity long bone bone defect treated with a microvascular fibula transfer in Helsinki University Central Hospital.

Exclusion Criteria:

* No upper extremity free fibular transfer

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Twenty patients with upper extremity long bone bone defect treated with a microvascular fibula transfer. Population aged below 90 years.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The long-term results are good | 10-20 years
  The long-term outcomes are assessed and good results gained.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand questionnaire | 10-20 years
  Assesses the function of the reconstructed limb
the 15-Dimensions health-related quality of life instrument | 10-20 years
  The 15-Dimensions assesses the health-related quality of life
Lower Extremity Functional Scale | 10-20 years
  Assesses the function of the donor site

CONTACTS AND LOCATIONS:
Overall Officials: Erkki J. Tukiainen, MD, PhD, Study Director — Helsinki University Central Hospital